CLINICAL TRIAL: NCT06169436
Title: 2014 Transizionali - Observational Study on the Occurrence of Relapses and on the Quality of Life in Patients Who Underwent Nephroureterectomy Surgery
Brief Title: Translational Cancer Observational Protocol
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Professor, IRCCS San Raffaele
Other Study IDs: 2014 - Transizionali
Record Dates: First submitted 2023-11-23; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma
Keywords: Upper Urinary Tract Urothelial Carcinoma; Nephroureterectomy surgery; Relapse; Quality of life; Diagnosis and Treatment strategies
MeSH Terms: conditions — Recurrence; Disease | interventions — Nephroureterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients with upper urinary tract urothelial cancer who underwent nephroureterectomy surgery
  Interventions: Procedure: Nephroureterectomy

INTERVENTIONS:
Procedure: Nephroureterectomy — Removal of cancer mass by urether and kidney complete resection.

SUMMARY:
Observational study on relapse occurrence and on the quality of life in patients who underwent nephroureterectomy surgery

DETAILED DESCRIPTION:
Monocentric prospective and retrospective observational study on the quality of life and on the pathological status in patients who underwent nephroureterectomy surgery. Oncological, psychological, sexual and quality of life-related data will be collected within a specifically created database that will allow us an easy and secure data extraction for the statistical analysis required by the clinical trial in terms of oncological relapse, clinical progression and improve the assistance and therapeutic strategy for each patient. Retrospective data for patients who underwent surgery between 1987 and today will be available in the form of clinical report stored in the hospital archives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Upper tract urothelial cancer diagnosis
* Indication to cancer removal through nephroureterectomy surgery
* Ability to read and sign the informed consent

Exclusion Criteria:

* Age < 18 years
* Absence of upper tract urothelial cancer
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper tract urothelial cancer who underwent nephroureterectomy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2014-07-17 (Actual); Primary Completion 2064-07-17 (Estimated); Study Completion 2064-07-17 (Estimated)

PRIMARY OUTCOMES:
Clinical progression data collection | 50 years
  Collection intended for the purpose of implementing diagnostic and therepautic strategies for the management of the disease in both the patient enrolled in the study and for future cases. Data will be collected in a dedicated internal database by means of medical records obtained during the patients' stay in the hospital and during follow up visits. The data collected includes anamnesis, data regarding surgery, laboratory exam and imaging exams.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No